CLINICAL TRIAL: NCT04047498
Title: Studying Stepping Control in Parkinson's Disease Using Alternating DBS
Brief Title: Alternating DBS for Stepping Control in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 230144
Record Dates: First submitted 2019-08-01; First posted 2019-08-06 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-07

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Masking Description: Participants and the UPDRS examiner are blinded to the stimulation condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Within-subjects comparison of constant and alternating DBS (Experimental)
  Interventions: Device: Alternating DBS

INTERVENTIONS:
Device: Alternating DBS — Constant DBS will be changed to DBS that is up- and downmodulated alternating between the left and right stimulation side.

SUMMARY:
Parkinson's disease (PD) is a disabling, progressive condition characterised by severe problems with movement for which medical treatment in the longer term can be unsatisfactory. Deep brain stimulation (DBS) is a treatment, which directly stimulates the nerve cells affected inside the brain to help overcome the difficulties with movement. Classically, DBS stimulates in a manner that is constant. Many patients develop severe problems with walking, so-called freezing of gait, which can be unresponsive to constant DBS. In this study the investigators will test if left-right alternating DBS helps to improve gait problems by potentially promoting left-right alternating up- and down-modulated brain activity, which was found during walking in a previous study. The investigators will test if alternating DBS improves the ability to adjust walking speed and to walk freely compared to constant DBS.

ELIGIBILITY:
Inclusion Criteria:

* PD patients with bilateral subthalamic nucleus DBS electrodes and stimulators implanted for at least 6 months
* Able to give consent.

Exclusion Criteria:

* Lack of capacity to consent
* Cognitive impairment/lack of capacity to perform experimental task. The investigators will additionally conduct a short (10 min) quantitative assessment of cognitive function using a validated test (MMSE). Patients with a score < 20 will be excluded from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Stepping control will be assessed as the ability to adjust the stepping speed (m/s) in each stimulation condition. | Immediate recording
  Stepping speed (m/s) will be assessed.
Stepping control will be assessed as the ability to limit the variance in stepping speed (m/s) in each stimulation condition. | Immediate recording
  Stepping variance (m/s) will be assessed.

SECONDARY OUTCOMES:
The investigators will test if patients automatically adjust to the stimulation rhythm | Immediate recording
  Stepping entrainment
The investigators will how well other motor symptoms including tremor, rigidity and bradykinesia are controlled with alternating DBS. | Immediate recording
  United Parkinsons Disease Rating Scale motor (Part III) scores will be compared between stimulation conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Brown, MD, Principal Investigator — University of Oxford
Locations (2):
- United Kingdom (2):
  - University College London Hospitals NHS Trust, London
  - University of Oxford, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be made available at https://data.mrc.ox.ac.uk/ once collected and fully analysed
Supporting Information: CSR
Time Frame: Anonymised data will be made available at https://data.mrc.ox.ac.uk/ once collected and fully analysed
Access Criteria: Please see https://data.mrc.ox.ac.uk/
URL: http://data.mrc.ox.ac.uk/

REFERENCES:
- [Background] Fischer P, Chen CC, Chang YJ, Yeh CH, Pogosyan A, Herz DM, Cheeran B, Green AL, Aziz TZ, Hyam J, Little S, Foltynie T, Limousin P, Zrinzo L, Hasegawa H, Samuel M, Ashkan K, Brown P, Tan H. Alternating Modulation of Subthalamic Nucleus Beta Oscillations during Stepping. J Neurosci. 2018 May 30;38(22):5111-5121. doi: 10.1523/JNEUROSCI.3596-17.2018. Epub 2018 May 14. PMID 29760182